CLINICAL TRIAL: NCT00113399
Title: A Phase III Trial for Locally Recurrent, Previously Irradiated Head and Neck Cancer: Concurrent Re-Irradiation and Chemotherapy Versus Chemotherapy Alone
Brief Title: Combination Chemotherapy With or Without Radiation Therapy in Treating Patients With Recurrent Head and Neck Cancer That Cannot Be Removed By Surgery
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated early due to low accrual.
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0421; CDR0000429480; ECOG-R0421
Record Dates: First submitted 2005-06-07; First posted 2005-06-08 (Estimated); Results first posted 2012-12-31 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-06

CONDITIONS: Head and Neck Cancer
Keywords: recurrent squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the oropharynx; recurrent metastatic squamous neck cancer with occult primary; recurrent lymphoepithelioma of the oropharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Filgrastim; Cisplatin; Docetaxel; Fluorouracil; Paclitaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radiotherapy and chemotherapy (Other): Radiotherapy/paclitaxel/cisplatin/filgrastim
  Interventions: Biological: filgrastim; Drug: cisplatin; Drug: paclitaxel; Radiation: radiation therapy
- Chemotherapy (Other): Cisplatin/fluorouracil/paclitaxel/docetaxel
  Interventions: Drug: cisplatin; Drug: docetaxel; Drug: fluorouracil; Drug: paclitaxel

INTERVENTIONS:
Biological: filgrastim
  Arms: Radiotherapy and chemotherapy
Drug: cisplatin
Drug: docetaxel
  Arms: Chemotherapy
Drug: fluorouracil
  Arms: Chemotherapy
Drug: paclitaxel
Radiation: radiation therapy
  Arms: Radiotherapy and chemotherapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Cisplatin and paclitaxel may make tumor cells more sensitive to radiation therapy. Giving more than one drug (combination chemotherapy) and giving them with radiation therapy may kill more tumor cells. It is not yet known whether giving radiation therapy together with combination chemotherapy is more effective than giving combination chemotherapy alone in treating head and neck cancer.

PURPOSE: This randomized phase III trial is studying radiation therapy and combination chemotherapy to see how well they work compared to combination chemotherapy alone in treating patients with recurrent head and neck cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare overall survival of patients with previously irradiated unresectable locally recurrent squamous cell carcinoma of the head and neck treated with radiotherapy, cisplatin, and paclitaxel vs cisplatin-based chemotherapy alone.

Secondary

* Compare progression-free survival of patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.
* Compare quality of life, functional/performance status, and quality-adjusted survival of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo radiotherapy twice daily and receive paclitaxel IV over 1 hour and cisplatin IV over 30 minutes once daily on days 1-5, 15-19, 29-33, and 43-47. Patients also receive filgrastim (G-CSF) subcutaneously once daily on days 6-13, 20-27, 34-41, and 48-55.
* Arm II: Patients receive 1 of the following cisplatin-based* regimens at the discretion of the treating physician:

  * Regimen 1: Patients receive cisplatin* IV over 1-2 hours on day 1 and fluorouracil IV continuously over 96 hours on days 1-4.
  * Regimen 2: Patients receive cisplatin* IV over 1-2 hours and paclitaxel IV over 3 hours on day 1.
  * Regimen 3: Patients receive cisplatin* IV over 1-2 hours and docetaxel IV over 1 hour on day 1.

NOTE: *Carboplatin may be substituted for cisplatin in patients with creatinine clearance < 50 mL/min or in patients who experience grade 2 or 3 neurotoxicity.

For all regimens, treatment repeats every 21 days for at least 6 courses in the absence of disease progression or unacceptable toxicity. Patients achieving complete response (CR) receive 2 additional courses beyond documentation of CR.

Quality of life is assessed at baseline and then at 3, 6, 12, 24, and 36 months.

After completion of study treatment, patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 240 patients (120 per treatment arm) will be accrued for this study within 5½ years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically* or cytologically* confirmed squamous cell carcinoma (SCC) of the oral cavity, oropharynx, hypopharynx, or larynx, including any of the following histologic variants:

  * Spindle cell carcinoma
  * Poorly differentiated keratin-positive carcinoma
  * Lymphoepithelioma NOTE: *Biopsy or primary tumor and/or fine needle aspiration of the metastatic lymph node required
* Original or second primary tumor

  * Recurrent neck metastases with unknown primary allowed
* Locally recurrent disease
* Measurable disease
* Unresectable disease

  * Attempted surgical resection allowed provided surgery was performed ≥ 3 months ago, wound is completely healed, and there is no sign of carotid exposure
* Must have had prior radiotherapy for SCC of the head and neck with > 75% of the present tumor volume in areas irradiated at doses ≥ 45 Gy but ≤ 75 Gy

  * Able to successfully re-irradiate the area of the gross tumor volume without exceeding lifetime spinal cord dose of 54 Gy as determined by physical examination and CT scan and/or MRI performed within the past 8 weeks
  * First recurrence occurred > 6 months after completion of radiotherapy

    * More than 1 recurrence allowed provided the above criteria for first recurrence has been met
* No primary tumor of the nasopharynx or salivary gland
* No distant metastases by history or physical examination, chest CT scan, and CT scan or MRI of the tumor site

  * Patients with equivocal pulmonary nodules are eligible provided the nodules are < 1 cm, can be safely biopsied, or are negative by positron emission tomography imaging
  * No circumferential tumor involvement of the carotid sheath by imaging unless prophylactic carotid stent is placed

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,800/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 8.0 g/dL (transfusion or other intervention allowed)

Hepatic

* AST or ALT < 2 times upper limit of normal (ULN)
* Bilirubin < 1.5 mg/dL
* No hepatic insufficiency resulting in clinical jaundice and/or coagulation defects

Renal

* Creatinine clearance > 50 mL/min
* Calcium < 11.5 mg/dL

Cardiovascular

* No New York Heart Association class III or IV heart disease
* No other symptomatic or uncontrolled cardiac disease

Pulmonary

* No chronic obstructive pulmonary disease exacerbation
* No other respiratory illness requiring hospitalization within the past 6 months or that would preclude study therapy

Immunologic

* No AIDS
* No prior allergic reaction to E. coli-derived products
* No acute bacterial or fungal infection requiring IV antibiotics

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 30 days after completion of study treatment
* No other invasive malignancy within the past 3 years except nonmelanoma skin cancer, carcinoma in situ of the breast, oral cavity, or cervix
* No pre-existing peripheral sensory neuropathy > grade 2
* No other severe active co-morbidity

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* At least 6 months since prior chemotherapy
* No prior systemic chemotherapy for recurrent SCC of the head and neck

  * Prior neoadjuvant, adjuvant, and/or concurrent chemotherapy and radiotherapy for initial SCC of the head and neck allowed

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* See Chemotherapy
* At least 6 months since prior radiotherapy

Surgery

* See Disease Characteristics

Other

* Prior cyclooxygenase-2 inhibitor or retinoids for chemoprevention allowed
* At least 6 months since prior epidermal growth factor receptor (EGFR) inhibitors or other targeted agents
* No prior EGFR inhibitors or other targeted agents for recurrent SCC of the head and neck
* No concurrent cimetidine or allopurinol (for patients on arm II, regimen 1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2005-04; Primary Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart J. Wong, MD, Principal Investigator — Medical College of Wisconsin
Locations (125):
- United States (125):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - St. Joseph's Mercy Cancer Center, Hot Springs, Arkansas
  - Auburn Radiation Oncology, Auburn, California
  - Radiation Oncology Centers - Cameron Park, Cameron Park, California
  - Mercy Cancer Center at Mercy San Juan Medical Center, Carmichael, California
  - Robert and Beverly Lewis Family Cancer Care Center at Pomona Valley Hospital Medical Center, Pomona, California
  - Radiation Oncology Center - Roseville, Roseville, California
  - Radiological Associates of Sacramento Medical Group, Incorporated, Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - Mercy General Hospital, Sacramento, California
  - Solano Radiation Oncology Center, Vacaville, California
  - Lynn Regional Cancer Center at Boca Raton Community Hospital - Main Center, Boca Raton, Florida
  - Michael & Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - Nancy N. and J. C. Lewis Cancer and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Saint James Hospital and Health Centers Comprehensive Cancer Institute - Olympia Fields, Olympia Fields, Illinois
  - Cancer Institute at St. John's Hospital, Springfield, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. John's Cancer Center at St. John's Medical Center, Anderson, Indiana
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Howard Community Hospital at Howard Regional Health System, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Reid Hospital & Health Care Services, Incorporated, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - MaineGeneral Medical Center - Waterville Campus, Waterville, Maine
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - Lakeland Cancer Care Center at Lakeland Hospital - St. Joseph, Saint Joseph, Michigan
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Missouri Regional Cancer Center at Southeast Missouri Hospital, Gape Girardeau, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Deaconess Billings Clinic - Downtown, Billings, Montana
  - Methodist Cancer Center at Methodist Hospital - Omaha, Omaha, Nebraska
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Kingsbury Center for Cancer Care at Cheshire Medical Center, Keene, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - J. Phillip Citta Regional Cancer Center at Community Medical Center, Toms River, New Jersey
  - Franklin & Edith Scarpa Regional Cancer Center at South Jersey Healthcare, Vineland, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - Long Island College Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Don Monti Comprehensive Cancer Center at North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Lenoir Memorial Cancer Center, Kinston, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Cancer Care Center at Medcenter One Hospital, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center, Bismarck, North Dakota
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Akron City Hospital, Akron, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Cancer Research UK Medical Oncology Unit at Churchill Hospital & Weatherall Institute of Molecular Medicine - Oxford, Salem, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - United States Air Force Medical Center - Wright-Patterson, Wright-Patterson AFB, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Mercy Fitzgerald Hospital, Darby, Pennsylvania
  - Alle-Kiski Medical Center, Natrona Heights, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - Cottonwood Hospital Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Latter Day Saints Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Norris Cotton Cancer Center - North, Saint Johnsbury, Vermont
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Community Memorial Hospital Cancer Care Center, Menomonee Falls, Wisconsin
  - Vince Lombardi Cancer Clinic at Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - All Saints Cancer Center at Wheaton Franciscan Healthcare, Racine, Wisconsin
  - University of Wisconcin Cancer Center at Aspirus Wausau Hospital, Wausau, Wisconsin
  - West Allis Memorial Hospital, West Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Re-irradiation Plus Concurrent Chemotherapy: Radiation Therapy on weeks 1, 3, 5, and 7; 1.5 Gy/fx, twice daily x 5 days, 40 fractions, for a total dose of 60 Gy; Chemotherapy (cisplatin/paclitaxel) on weeks 1, 3, 5, and 7 G-CSF on weeks 2, 4, 6, and 8. [Data is reported for eligible patients with adverse event information, which is 6 patients.]
- Chemotherapy Alone: Select from one of the three standard chemotherapy regimens:
  cisplatin/5-FU; cisplatin/paclitaxel; cisplatin/docetaxel. [Data is reported for eligible patients with adverse event information, which is 7 patients.]
Period: Overall Study
Arm/Group | Re-irradiation Plus Concurrent Chemotherapy | Chemotherapy Alone
Started | 7 | 8
Completed | 5 | 3
Not Completed | 2 | 5
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Complete Response | 0 | 1
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Re-irradiation Plus Concurrent Chemotherapy: Radiation Therapy on weeks 1, 3, 5, and 7 1.5 Gy/fx, twice daily x 5 days, 40 fractions, for a total dose of 60 Gy; Chemotherapy (cisplatin/paclitaxel) on weeks 1, 3, 5, and 7 G-CSF on weeks 2, 4, 6, and 8. [Data is reported for eligible patients with on-study information, which is 6 patients.]
- Chemotherapy Alone: Select from one of the three standard chemotherapy regimens:
  cisplatin/5-FU; cisplatin/paclitaxel; cisplatin/docetaxel. [Data is reported for eligible patients with on-study information, which is 7 patients.]
- Total: Total of all reporting groups
Arm/Group | Re-irradiation Plus Concurrent Chemotherapy | Chemotherapy Alone | Total
Number analyzed (Participants) | 6 | 7 | 13
Age Continuous [Median (Full Range); unit: years] | 56 [44 to 80] | 57 [48 to 68] | 57 [44 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Time Frame: Date of death or last follow-up
Population: This study terminated early with 15 subjects out of 240 subjects accrued, therefore no analyses were performed.
Groups:
- Re-irradiation Plus Concurrent Chemotherapy: Radiation Therapy on weeks 1, 3, 5, and 7 1.5 Gy/fx, twice daily x 5 days, 40 fractions, for a total dose of 60 Gy Chemotherapy (cisplatin/paclitaxel) on weeks 1, 3, 5, and 7 G-CSF on weeks 2, 4, 6, and 8
- Chemotherapy Alone: Select from one of the three standard chemotherapy regimens:
  cisplatin/5-FU; cisplatin/paclitaxel; cisplatin/docetaxel
Arm/Group | Re-irradiation Plus Concurrent Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Per the protocol, toxicity data was collected via CTCAE 3.0, then mapped to CTCAE 4.0 for reporting on this website. Subjects experiencing > 1 of a given SAE are counted only once for that SAE. Subjects experiencing > 1 of a given "Other (Not Including Serious)" AE are counted only once for that "Other (Not Including Serious)" AE.
Arm/Group | Re-irradiation Plus Concurrent Chemotherapy | Chemotherapy Alone
Serious Adverse Events (participants affected / at risk) | 4/6 | 4/7
Other Adverse Events (participants affected / at risk) | 6/6 | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Re-irradiation Plus Concurrent Chemotherapy (N=6) | Chemotherapy Alone (N=7)
Cardiac disorders - Other (Cardiac disorders) | 0 | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Allergic reaction (Immune system disorders) | 0 | 1
Bronchial infection (Infections and infestations) | 0 | 1
Infections and infestations - Other (Infections and infestations) | 2 | 0
Neutrophil count decreased (Investigations) | 1 | 1
White blood cell decreased (Investigations) | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypotension (Vascular disorders) | 1 | 2
Thromboembolic event (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Re-irradiation Plus Concurrent Chemotherapy (N=6) | Chemotherapy Alone (N=7)
Anemia (Blood and lymphatic system disorders) | 6 | 5
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 0 | 1
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 1
Hearing impaired (Ear and labyrinth disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 3
Diarrhea (Gastrointestinal disorders) | 1 | 2
Dry mouth (Gastrointestinal disorders) | 4 | 1
Dysphagia (Gastrointestinal disorders) | 3 | 2
Esophageal pain (Gastrointestinal disorders) | 1 | 1
Esophagitis (Gastrointestinal disorders) | 3 | 0
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 3 | 5
Oral cavity fistula (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 2 | 5
Edema face (General disorders) | 1 | 0
Fatigue (General disorders) | 5 | 4
Fever (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Infections and infestations - Other (Infections and infestations) | 1 | 1
Lung infection (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 0 | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 2 | 0
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 1
Alanine aminotransferase increased (Investigations) | 2 | 0
Alkaline phosphatase increased (Investigations) | 5 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 0
Creatinine increased (Investigations) | 1 | 2
Investigations - Other (Investigations) | 1 | 1
Lymphocyte count decreased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 2 | 2
Platelet count decreased (Investigations) | 4 | 3
Weight loss (Investigations) | 3 | 1
White blood cell decreased (Investigations) | 5 | 2
Anorexia (Metabolism and nutrition disorders) | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 5 | 4
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 3 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 5 | 4
Hypoglycemia (Metabolism and nutrition disorders) | 3 | 2
Hypokalemia (Metabolism and nutrition disorders) | 3 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 3 | 1
Hyponatremia (Metabolism and nutrition disorders) | 5 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 0
Iron overload (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 2
Dysgeusia (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 4
Anxiety (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin induration (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 1
Hot flashes (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
This study terminated early with 15 subjects out of 240 subjects accrued, therefore no analysis was performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No